CLINICAL TRIAL: NCT01918345
Title: Avoiding Diabetes After Pregancy Trial in Moms (ADAPT-M): Pilot, Feasibility and Effectiveness Phases
Brief Title: Avoiding Diabetes After Pregnancy Trial in Moms
Acronym: ADAPT-M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: The Lawson Foundation (Other); Diabetes Canada (Other); Unity Health Toronto (Other); Sunnybrook Health Sciences Centre (Other); Mount Sinai Hospital, Canada (Other); Michael Garron Hospital (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Scarborough Rouge Hospital (Other); J.P. Bickell Foundation (Unknown)
Responsible Party: Principal Investigator, Lorraine Lipscombe, Endocrinologist, Research Scientist, Women's College Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: ADAPT2013
Record Dates: First submitted 2013-07-31; First posted 2013-08-07 (Estimated); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Diabetes
Keywords: Diabetes; Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes, gestational; Prevention & control; Postpartum Period; Mothers; Diet; Diabetic Diet; Exercise; Life Style; Motivation; Health Behavior; Insulin-Secreting Cells; Randomized Controlled Trial; Clinical Trial; Pilot Projects; Feasibility Studies
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes, Gestational; Motor Activity; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard Care (Control) (No Intervention): This group will receive a one-on-one counseling session during one visit with a Certified Diabetes Educator (CDE), who will provide standard advice on diabetes prevention and healthy lifestyle. They will receive a booklet on exercise and healthy diet as per current Canadian guidelines for healthy eating. This group will also receive a check-in telephone call from the Study Coordinator, half-way through the study. This group will not receive motivational interviewing, health coaching on low GI diet and/or exercise, or additional telephone follow-up.
- Diet & Physical Activity Program with Health Coach (Experimental): Participants assigned to this arm will receive a combination of the home-based physical activity program with health coach and the home-based low-GI diet program with health coach, as described in the respective individual arms. The Health Coach for this group will be a CDE.
  Interventions: Behavioral: Home-based Physical Activity Program with Health Coach; Behavioral: Home-based Low-GI Diet Program with Health Coach
- Physical Activity Program with Health Coach (Experimental): Participants will be counseled to follow physical activity recommendations for Canadians, which is at least 150 minutes of moderate physical activity per week. Participants will be asked to participate in aerobic, strength training and stretching activities. Health Coaches will use motivational interviewing, goal-setting and problem solving to assist participants in meeting their physical activity goals. More participants will be randomized to this group and the participants will either have CDE or a Registered Kinesiologist (R. Kin) as their health coach.
  Interventions: Behavioral: Home-based Physical Activity Program with Health Coach
- Diet Program with Health Coach (Experimental): Participants will be counseled to follow recommendations for Canadians on healthy eating (Canada's Food Guide and Space on Your Plate. Low GI education will be layered on top of Canada's Food Guide recommendations. The goal for participants in the diet group is to lower their dietary GI by 8-10 units. Health Coaches will use motivational interviewing, goal-setting and problem solving to assist participants in meeting their dietary and low GI goals. The health coach for this group will be a CDE.
  Interventions: Behavioral: Home-based Low-GI Diet Program with Health Coach

INTERVENTIONS:
Behavioral: Home-based Physical Activity Program with Health Coach — This arm will receive either a trained CDE or R. Kin as a health coach and a home-based physical activity program for 6 months. Health coaches will provide one-on-one motivational interviewing (MI) and goal-setting, and will account for baseline fitness, resources, childcare, and breastfeeding, to be undertaken at participants' homes or in their communities. Prescriptions will be based on minimum recommendations for moderate-intensity exercise for postpartum women. Participants will maintain at least 150 min/week of moderate activity at a target heart rate of 30-80% with a perceived exertion of 12-15 on the Borg Scale. They will also be counseled on resistance training and pelvic floor exercises. They will receive regular telephone-based coaching to advance goals. Phone-calls will be administered on a weekly basis during weeks 2-8 of the intervention, biweekly basis on weeks 10-12, and monthly basis on weeks 16-24.
  Arms: Diet & Physical Activity Program with Health Coach; Physical Activity Program with Health Coach
Behavioral: Home-based Low-GI Diet Program with Health Coach — This arm will receive a trained CDE health coach and a home-based low-GI diet program for 6 months. Health coaches will provide baseline education during a one-on-one visit and use MI to introduce the dietary intervention. Low GI education will be layered on top of current standard care, which asks women to consume a diet comprised of 45-65% carbohydrates (25 g of dietary fibre), 10-30% protein, and 25-35% fat. As per standard care at the DEPs, this intake will be divided into 3 meals and 2 to 4 snacks. Resources for women will include a low GI dietary food substitution list, a recipe booklet, and a tip sheet on how to lower dietary GI. Women will receive regular telephone-based coaching to advance goals. Phone-calls will be administered on a weekly basis during weeks 2-8 of the intervention, biweekly basis on weeks 10-12, and monthly basis on weeks 16-24.
  Arms: Diet & Physical Activity Program with Health Coach; Diet Program with Health Coach

SUMMARY:
Mothers with previous gestational diabetes mellitus (GDM) represent a population at higher risk of future Type 2 diabetes mellitus (T2DM), which is preventable through lifestyle modification. Yet, no formal prevention programs exist for this population. The postpartum period is a particularly vulnerable period for weight gain and unhealthy lifestyle in new mothers due to their competing demands of childcare and breastfeeding. This important time period may thus represent a 'window of opportunity' for women with previous GDM, whereby interventions to improve their lifestyle can be offered. Eligible women will be recruited during pregnancy from four hospitals and invited to participate in a home-based lifestyle intervention program starting from three to six months postpartum. This pilot study will investigate the feasibility and effectiveness of a physical activity and diet intervention. It will also explore the relationship between behaviour change and metabolic markers of T2DM in this high-risk population. Investigators hypothesize that the ADAPT-M program will be feasible and will be associated with an improvement in metabolic T2DM markers, as well as a high rate of satisfaction, adherence, and effectiveness.

DETAILED DESCRIPTION:
Women diagnosed with gestational diabetes mellitus (GDM) are a readily identifiable population at high risk for type 2 diabetes (T2DM) to whom preventive interventions can be offered. There is evidence that T2DM can be prevented with lifestyle modification in older high-risk risk groups. However, preventive trials for women with recent GDM have had limited success in preventing T2DM, in part because they have failed to produce significant behaviour change. New mothers are a unique population with many competing demands and barriers to behaviour change. Home-based health coaching programs may be more effective in women with recent GDM, as they provide greater flexibility, goal-setting, and frequent follow-up, and have been associated with greater adherence and weight loss. Low glycemic-index diets are also associated with greater adherence and improved glycemia, but data are lacking in women with recent GDM.

The ADAPT-M (Avoiding Diabetes after Pregnancy Trial in moms) study will address these gaps by evaluating a home-based exercise and diet intervention that has been designed specifically for new mothers with recent GDM. An internationally renowned team of investigators and collaborators was brought together to create this intervention. This trial has been carefully designed based on our previous work, an extensive literature review, and the input from co-investigators with expertise in diabetes research, gestational diabetes, prenatal and postpartum care, diabetes education programs, home-based exercise coaching, nutrition and diet interventions, and clinical trials. Investigators will work closely with the Clinical Trials Unit of the Applied Health Research Centre (AHRC) of University of Toronto to develop, implement, and evaluate this trial.

This study is important because it addresses a crucial missed opportunity for diabetes prevention in a well-defined, high-risk population. This intervention is unique because it has been specifically tailored to optimize behaviour change by meeting the needs of new mothers. The findings from this study will have implications for diabetes caregivers, policy-makers, and researchers. This work will benefit women with prior GDM and their families by offering a much-needed effective and sustainable program aimed at reducing their risk of diabetes and improving long-term health.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Physician-diagnosed Gestational Diabetes Mellitus (GDM) during most recent pregnancy based on Canadian Diabetes Association (CDA) diagnostic criteria
* 3-6 months postpartum after a GDM pregnancy
* During GDM pregnancy, followed by a Diabetes In Pregnancy clinic at one of study sites (i.e. Sunnybrook Health Sciences Centre, Mount Sinai Hospital, St. Michael's Hospital, Toronto East General Hospital)
* English-speaking

Exclusion Criteria:

* Current diabetes (Type I or Type II) and/or treatment with any anti-diabetic therapy
* Any major illness that may interfere with participation
* Any obstetrical or fetal complication that may interfere with participation
* Involvement in any other clinical trial requiring drug therapy
* History of cardiovascular disease or ECG abnormalities on stress echo cardiogram
* New pregnancy within postpartum period
* Any illness affecting carbohydrate digestion and/or metabolism including kidney disease, hepatitis, HIV/AIDS, celiac disease
* Any other factor likely to limit study adherence, in the opinion of the principal investigator
* (For the Effectiveness Phase ONLY) Participation in the Pilot Phase of the ADAPT-M Study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2014-07; Primary Completion 2022-10 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
For the Pilot Phase: Change in baseline-adjusted pancreatic beta-cell function | Assessed at week 1 (baseline) and week 24 (study end) of intervention
  Beta-cell function will be measured using the Insulin Secretion Sensitivity Index 2 (ISSI-2), which is an established oral glucose tolerance test (OGTT)-based measure of beta-cell function that has been validated against the disposition index from intravenous glucose tolerance test (ivGTT) and has been used in previous clinical trials. ISSI-2 is the product of insulin secretion [the ratio of area under-the-insulin-curve (AUCins) to area-under-the-glucose curve (AUCgluc)] and insulin sensitivity measured by the Matsuda index:
  ISSI-2 = (AUCins / AUCgluc) × [10000 / √(Fglu × Fins × Mglu × Mins)]
  Where Fglu = fasting glucose; Fins = fasting insulin; Mglu = mean glucose; Mins = mean insulin
  These measures will be calculated using the glucose and insulin values at baseline, and at 60 and 120 minutes following a 75-gram oral glucose load.
For the Effectiveness Phase: Change in baseline-adjusted weight | Assessed at week 1 (baseline) and week 24 (study end) of intervention
  For the effectiveness phase weight is now the primary outcome and change in baseline-adjusted pancreatic beta-cell function a secondary outcome. Weight in kilograms (kg) will be measured using a medical grade scale at the baseline and final health assessment.. We will also measure height in metres (m) using a medical grade stadiometer to calculate body-mass index (BMI, kg/m2). We will analyze the weight and height outcomes as continuous variables. We will then categorize BMI as under/normal weight (< 25 kg/m2), overweight (25.1-29.9 kg/m2), and obese (≥ 25 kg/m2). Finally, we will also calculate the proportion of participants who return to their pre-pregnancy weight or less, based on self-reported pre-pregnancy weight.

SECONDARY OUTCOMES:
Feasibility | Assessed at week 12 (mid-study) and 24 (study end) of intervention
  Feasibility measures will include recruitment, pre- and post-randomization attrition, adherence and follow-up rates, and symptoms, side effects, and satisfaction of the interventions. Adherence to exercise will be assessed with the International Physical Activity Questionnaire (IPAQ), physical activity records and accelerometer administered/worn at baseline, mid-study (week 12 of intervention) and follow-up, which estimates whether activity guidelines are met. Participant log books will be reviewed to assess diet and exercise adherence. Optimal adherence will be defined as meeting activity guidelines or consuming low GI foods at least 60% of the time for the exercise and diet arms respectively. Safety of interventions will also be assessed based on self-reported symptoms and side effects during telephone follow-up and at study end.
  Participants will also complete questionnaires on satisfaction of the education and interventions throughout the study and at study end.

OTHER OUTCOMES:
Behaviour change | Assessed at week 1 (baseline) and week 24 (study end) of intervention
  Exercise capacity: The primary endpoint for the exercise intervention will be baseline-adjusted exercise capacity at study end based on peak oxygen consumption (VO2max) from the graded exercise treadmill test. Change in metabolic equivalents (METs) and percent age-predicted fitness will also be calculated based on the Bruce protocol:
  % age-predicted fitness = (100×observed MET)/age-predicted MET, where MET = VO2max / 3.5
  Diet GI: The primary endpoint for the low GI diet intervention will be baseline-adjusted diet GI, which will be calculated using a three-day diet record using the following validated formula:
  Dietary GI = [ΣC×F×GI]/[ΣC×F]
  Where C=quantity of carbohydrate in age-specific portion of food; F=frequency of consumption/day; GI = GI of the food with glucose as the reference (GI=100).

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine L Lipscombe, MD, MSc, FRCPC, Principal Investigator — Women's College Hospital
Locations (5):
- Canada (5):
  - Scarborough Health Network, Scarborough Village, Ontario
  - Michael Garron Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario